CLINICAL TRIAL: NCT03866551
Title: Reprieve Cardiovascular System for the Treatment of Subjects With Acute Decompensated Heart Failure
Brief Title: Reprieve ADHF EFS IDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CardioRenal Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCV-0001
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Congestive Heart Failure
Keywords: Acute Heart Failure; Decompensated Heart Failure; Heart Failure Treatment; Heart Failure Management Fluid Overload; Diuresis
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Interventional Arm (Experimental): The initial phase of the study will utilize the Reprieve Cardiovascular System to support a treatment algorithm that maximizes diuretic administration while carefully monitoring patient physiologic and hemodynamic status to ensure safe decongestion.
  Interventions: Device: Reprieve Cardiovascular System

INTERVENTIONS:
Device: Reprieve Cardiovascular System — The Reprieve Cardiovascular System (RCS) shall be utilized to maximize fluid removal over a maximum duration of 72 hours.

SUMMARY:
This is a prospective, single arm, early feasibility study (EFS) designed to evaluate the safety and device performance of The RenalGuard System in the management of patients admitted with signs and symptoms of congestive heart failure who require diuresis for the treatment of volume overload.

DETAILED DESCRIPTION:
This is a prospective, single arm, early feasibility study (EFS) designed to evaluate the safety and device performance of The Reprieve System in the management of patients admitted with signs and symptoms of congestive heart failure who require diuresis for the treatment of volume overload. Subjects will be referred by their physician if he/she feels that the subject could benefit from observed diuresis in a hospital setting.

The device being utilized is called The Reprieve System (The System). By default, The System infuses a volume of hydration fluid equal to the volume of urine output. This is known as matched hydration. In addition, the clinician has the ability to adjust the matched setting such that RenalGuard can infuse hydration fluid to achieve a positive fluid balance (e.g. +100 ml/hr.) or a negative fluid balance (e.g. -100 ml/hr.). The purpose of this balanced fluid replacement is to prevent hypovolemia that may lead to hypotension and vital organ dysfunction, or fluid overload that may lead to shortness of breath in subjects in whom high urine output is desired.

All patients will be treated with The Reprieve System for up to 72-hours, at the investigators discretion. They will be followed for 30 days post discharge. The protocol will enroll up to 40 subjects to develop the clinical algorithm required to optimally and safely perform removal of volume. The study will be conducted in up to 5 sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for participation in the study must meet all of the following inclusion criteria. It is anticipated that this population will include Medicare beneficiaries as the patient population is generally greater than 65 years of age:

  1. Patients > 18 years of age
  2. Hospitalized with an episode of acute decompensated heart failure based on testing positive with at least two of the following:

     1. Persistent dyspnea at rest or with minimal exertion despite standard background therapy for acute heart failure including treatment with furosemide;
     2. Edema > +1 on a 0-3+ scale, indicating indentation of skin with mild digital pressure that requires 10 or more seconds to resolve in any dependent area including extremities or sacral region;
     3. Radiological evidence of pulmonary congestion on a chest X-ray (if an appropriate chest computerized tomography scan is done; the X-ray need not be performed);
  3. Systolic BP ≥ 90 mg Hg and ≤ 180 mm Hg without the need for inotropes or vasopressors at the time of enrollment.
  4. Currently receiving loop diuretics (e.g. bumetanide, torsemide, furosemide) as home therapy for a minimum of 6 months prior to admission.
  5. Capable of giving written informed consent, willing to comply with study procedures
  6. Females of childbearing age should use adequate contraceptives.

Exclusion Criteria:

Candidates for participation will be ineligible for the study if any of the following exclusion criteria apply:

1. Acute or suspected acute myocardial infarction (AMI) or troponin levels > 3X the upper limit of normal at the institution's local laboratory.
2. Inability to place Foley catheter or IV catheter.
3. Dyspnea due to non-cardiac causes (i.e. severe chronic obstructive pulmonary disease, bronchitis, pneumonia) which may interfere with the ability to interpret the primary cause of dyspnea.
4. Cardiogenic shock.
5. Acute systemic infection.
6. Sustained heart rate > 130 bpm.
7. AHF due to significant arrhythmias, which include any of the following: sustained ventricular tachycardia or atrial fibrillation/ flutter with sustained ventricular response of >130 beats per minute; or bradycardia with sustained ventricular rate <45 beats per minute without the use of a pacemaker.
8. Patients with hemoglobin < 8 g/dl, or a history of blood transfusion within the 14 days prior to screening, or active life-threatening GI bleeding.
9. Impaired renal function based upon a GFR of <20 ml/min/1.73m2 calculated using the aMDRD equation.
10. Current or planned ultrafiltration, hemofiltration, or dialysis.
11. Known hepatic impairment (as evidenced by total bilirubin >3mg/dL, or increased ammonia levels, if performed) or history of cirrhosis with evidence of portal hypertension such as varices.
12. Significant, uncorrected, left ventricular outflow obstruction, such as obstructive hypertrophic cardiomyopathy; or severe aortic stenosis (i.e., aortic valve area <1.0 cm2 or mean gradient >40mmHg on prior or current echocardiogram); or severe mitral stenosis.
13. Any major solid organ transplant recipient or planned/anticipated organ transplant within 1 year.
14. Major surgery or Major neurologic event, including cerebrovascular events in the 30 days.
15. Acute myocarditis or hypertrophic obstructive, restrictive, or constrictive cardiomyopathy (Note: restrictive mitral filling patterns noted on Transthoracic Echocardiography Assessment of diastolic function is not an exclusion).
16. Severe aortic insufficiency or severe mitral regurgitation for which surgical or percutaneous intervention is indicated.
17. Documented history of restrictive amyloid myocardiopathy, OR acute myocarditis or hypertrophic obstructive, restrictive, or constrictive cardiomyopathy (Note: restrictive mitral filling patterns noted on Transthoracic Echocardiography Assessment of diastolic function is not an exclusion).
18. Current (within 2 hours prior to enrollment) or planned (through the completion of the Reprieve Cardiovascular System use) treatment with any IV vasoactive therapies, including vasodilators (including nesiritide), positive inotropic agents and vasopressors, or mechanical support (i.e. endotracheal intubation, mechanical ventilation; intra-aortic balloon pump or any ventricular assist device; with the exception of IV furosemide (or equivalent diuretic), IV renal dopamine <5mcg/kg/min, or IV nitrates at a dose of ≤0.1mg/kg/hour if the patient has a systolic BP >150mmHg at the start of screening.
19. Use of any investigational drugs within 30 days prior to screening.
20. Inability to follow instructions or comply with follow-up procedures.
21. Pregnant females or females anticipating pregnancy during study period.
22. Patients currently enrolled in another interventional clinical study.
23. Other concomitant disease or condition that may put the patient at risk or influence study results in the investigator's opinion, or that the investigator deems unsuitable for the study, including drug or alcohol abuse or psychiatric, behavioral or cognitive disorders, sufficient to interfere with the patient's ability to understand and comply with the protocol instructions or follow-up procedures.
24. Anuria
25. Established sensitivity to furosemide
26. Significant hypokalemia (e.g., <3.0 mEq/L)
27. Significant hypomagnesemia (e.g., <1.8 mg/dL)
28. Significant hypocalcemia (e.g., total, <7.5 mg/dL; ionized, <4.0 mg/dL)
29. Use of nephrotoxic agents (this criterion should not prevent use of nephrotoxic agents during therapy if deemed to be clinically necessary)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
72 hour fluid removal | 72 hours
  The ability to remove at least 5L of fluid and/or demonstrate clinical decongestion at completion of treatment with the Reprieve Cardiovascular System (maximum 72 hours on treatment with RCS).